CLINICAL TRIAL: NCT07153575
Title: Comparison of the Postoperative Analgesic Effectiveness of Suprainguinal Fascia Iliaca Block (SFIB) and Pericapsular Nerve Block (PENG) in Hip Arthroplasty
Brief Title: Postoperative Analgesia in Hip Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Fatih Ugun, Assistant Professor, MD, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023/142
Record Dates: First submitted 2025-05-03; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hip Fractures; Post Operative Pain; Postoperative Nausea and Vomiting
Keywords: Hip Arthroplasty; Postoperative analgesia; Suprainguinal fascia iliaca block; Pericapsular nerve group block
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suprainguinal fascia iliaca block (Active Comparator): The ultrasound-guided suprainguinal fascia iliaca block (SFIB) procedure was first described by Hebbard et al. in 2011. It is a prevalent regional anesthesia technique employed in surgical procedures involving the hip joint and femur. Local anesthetics are administered in close proximity to the fascia iliaca. The primary objective is to obstruct the femoral, obturator and lateral femoral cutaneous nerve in a simultaneous manner. In clinical practice, it is a safe and simple alternative to lumbar plexus blocks and femoral blocks. A 30-ml solution of 0.25% bupivacaine was injected between the iliac muscle and the iliac fascia. The bupivacaine dosage administered in the study was standardized for the groups by employing equal concentrations and volumes.
  Interventions: Procedure: suprainguinal fascia iliaca block
- Pericapsular nerve group block (Active Comparator): In pericapsular nerve group (PENG) block the local anesthetic agent is injected into the musculofascial plane between the psoas muscle tendon and the pubic ramus. The primary objective of this technique is to obstruct the genicular branches of the femoral, obturator, and accessory obturator which innervate the hip capsule. Therefore, a comparison with the SFIB was undertaken. A 30-ml block of 0.25% bupivacaine solution was injected between the pubic ramus and the iliopsoas muscle tendon. The bupivacaine dosage administered in the study was standardized for the groups by employing equal concentrations and volumes.
  Interventions: Procedure: Pericapsular nerve group (PENG) block

INTERVENTIONS:
Procedure: suprainguinal fascia iliaca block — The ultrasound-guided suprainguinal fascia iliaca block (SFIB) procedure was first described by Hebbard et al. in 2011. It is a prevalent regional anesthesia technique employed in surgical procedures involving the hip joint and femur. Local anesthetics are administered in close proximity to the fascia iliaca. The primary objective is to obstruct the femoral, obturator and lateral femoral cutaneous nerve in a simultaneous manner. In clinical practice, it is a safe and simple alternative to lumbar plexus blocks and femoral blocks. A 30-ml solution of 0.25% bupivacaine was injected between the iliac muscle and the iliac fascia. The bupivacaine dosage administered in the study was standardized for the groups by employing equal concentrations and volumes.
  Arms: Suprainguinal fascia iliaca block
Procedure: Pericapsular nerve group (PENG) block — In pericapsular nerve group (PENG) block the local anesthetic agent is injected into the musculofascial plane between the psoas muscle tendon and the pubic ramus. The primary objective of this technique is to obstruct the genicular branches of the femoral, obturator, and accessory obturator which innervate the hip capsule. Therefore, a comparison with the SFIB was undertaken. A 30-ml block of 0.25% bupivacaine solution was injected between the pubic ramus and the iliopsoas muscle tendon. The bupivacaine dosage administered in the study was standardized for the groups by employing equal concentrations and volumes.
  Arms: Pericapsular nerve group block

SUMMARY:
The goal of this clinical trial is to compare analgesic effectiveness of two blocks in hip arthroplasty. The main question that aim to answer is;

-Which block is more efficient? Researchers will compare suprainguinal fascia iliaca block with perineural nerve group block.

Participants will randomized and one of the blocks will be applied.

DETAILED DESCRIPTION:
Postoperative pain and analgesia in hip surgery is an important issue for early mobilization and length of hospital stay. The patient population is usually elderly. Prolonged hospital stay may cause thromboembolic complications due to delayed mobilization, psychiatric conditions such as delirium, and many undesirable conditions caused by pain such as chronicisation of acute pain. There are neuraxial analgesia, regional analgesia and multimodal analgesia regimens that are used together to prevent postoperative pain and to prevent these undesirable conditions caused by pain. Suprainguinal fascia iliaca block and pericapsular nerve group blocks are two of those. With performing these blocks, we will obtain postoperative analgesia and avoid postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer patients undergoing hip arthroplasty
* Voluntary patient to undergo elective operation under regional anaesthesia
* ASA I-II-III
* BMI≤35 kg/m²

Exclusion Criteria:

* Obstacles to the application of regional anaesthesia
* Local Anaesthetic Allergy
* Coagulopathy
* Psychiatric disorders and medication
* Hematological/Oncological disease
* Severe organ failure
* Multiple bone fractures
* Alcohol/Drug addiction
* Used analgesic medication up to 12 hours before surgery
* Infection at the Block Application Site
* Mental Deficiency
* Morbidly obese patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
To compare the postoperative analgesic efficacy of SFIB and PENG block | 24 hours
  Calculating total morphine consumption over 24 hours in patients by using patient controlled analgesia pump.

SECONDARY OUTCOMES:
Postoperative analgesia scores | 24 hours
  Detecting postoperative analgesia scores during rest and movement by using Numerical Rating Scale (NRS) scores. The scale ranges from 0 - 10. Zero represents no pain, while 10 represents the worst possible pain.
Assessment of nausea and vomiting incidence | 24 hours
  The incidence of nausea and vomiting was examined at 1, 3, 6, 12, 18, and 24 hours post-intervention. The data were analyzed across groups using a 4-point categorical scoring system, with the following definitions: No nausea: 0; Mild: 1; Moderate: 2; Severe: 3.

OTHER OUTCOMES:
Satisfaction levels | 24 hour
  An assessment was also conducted to determine the subjects' satisfaction levels using the Quality of Recovery-15T (QoR-15T) survey at 24th hour. This scale provides a score ranging from 0 to150, with a high score indicating a good quality of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Ugün, M.D., Principal Investigator — Balikesir University
Locations (1):
- Balikesir University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD throughout the trial will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 1 year after the publication of results
Access Criteria: All study data and analysis stages will be shared with interested researchers 1 year after the study is published.

REFERENCES:
- See also: Ultrasound-guided, direct suprainguinal injection for fascia iliaca block for total hip arthroplasty: A retrospective study — https://pubmed.ncbi.nlm.nih.gov/34046456/
- See also: Comparison of conventional infrainguinal versus modified proximal suprainguinal approach of Fascia Iliaca Compartment Block for postoperative analgesia in Total Hip Arthroplasty. A prospective randomized study — https://pubmed.ncbi.nlm.nih.gov/26767235/
- See also: Comparative evaluation of femoral nerve block and intravenous fentanyl for positioning during spinal anaesthesia in surgery of femur fracture — https://pubmed.ncbi.nlm.nih.gov/25624533/
- See also: Comparison of pericapsular nerve group (PENG) block with fascia iliaca compartment block (FICB) for pain control in hip fractures: A double-blind prospective randomized controlled clinical trial — https://pubmed.ncbi.nlm.nih.gov/34715388/
- See also: Ultrasound guided Fascia Iliaca Block versus Pericapsular Nerve Group for Postoperative Analgesia Prior to Spinal Anaesthesia for Hip Surgeries — https://doi.org/10.53730/ijhs.v6nS4.6117
- See also: Effectiveness of perineural administration of dexamethasone with lidocaine on onset time of sensory block and early postoperative analgesia in axillary brachial plexus block: a prospective cohort study, Ethiopia — https://pubmed.ncbi.nlm.nih.gov/38463067/
- See also: Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty — https://pubmed.ncbi.nlm.nih.gov/34290085/
- See also: Comparison of the efficacy of pericapsular nerve group block (PENG) block versus suprainguinal fascia iliaca block (SFIB) in total hip arthroplasty: A randomized control trial — https://pubmed.ncbi.nlm.nih.gov/37303868/
- See also: Effect of pericapsular nerve group block and suprainguinal fascia iliaca block on postoperative analgesia and stress response in elderly patients undergoing hip arthroplasty: a prospective randomized controlled double-blind trial — https://pubmed.ncbi.nlm.nih.gov/38956469/
- See also: Effects of Perioperative Fascia Iliaca Compartment Block on Postoperative Pain and Hip Function in Elderly Patients With Hip Fracture — https://pubmed.ncbi.nlm.nih.gov/35450298/